CLINICAL TRIAL: NCT01852799
Title: A Phase 2, Multicenter, Single Arm Study to Evaluate the Effect of PAD Followed by Autologous Stem-cell Transplantation(ASCT) on the Concentrations of Bone Metabolites in Patients With Newly Diagnosed Multiple Myeloma(MM)
Brief Title: A Study of PAD Followed by Autologous Stem Cell Transplantation (ASCT) to Treat Newly Diagnosed Multiple Myeloma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Shanghai Changzheng Hospital (Other)
Responsible Party: Principal Investigator, Jian Hou, Chief Physician, Professor of Shanghai Changzheng Hospital, Shanghai Changzheng Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 26866138MMY2074
Record Dates: First submitted 2013-04-28; First posted 2013-05-14 (Estimated); Results first posted 2018-08-10 (Actual); Last update posted 2018-08-10 (Actual); Status verified 2017-11

CONDITIONS: Multiple Myeloma
Keywords: Multiple myeloma; PAD; ASCT; Bone metabolites; Bone marker
MeSH Terms: conditions — Multiple Myeloma | interventions — Neoadjuvant Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- PAD Followed by ASCT (Experimental): Drug: Bortezomib, Adriamycin (Doxorubicin) /Epidoxorubicin(EPI), Dexamethasone.
  After received induction therapy, patients will proceed to receive ASCT based on the willing of the patients and the decision of the investigators.
  Interventions: Drug: PAD Followed by ASCT

INTERVENTIONS:
Drug: PAD Followed by ASCT — Drug: Bortezomib, Bortezomib (1.3mg/m2, iv, on day 1, 4, 8, 11, of each 28 day cycle)
  Drug: Adriamycin (Doxorubicin) /EPI, Adriamycin (Doxorubicin) (9 mg/m2, iv, on days 1-4 of each 28 day cycle) or EPI (15mg/m2, iv, on days 1-4 of each 28 day cycle)
  Drug: Dexamethasone, Dexamethasone (20mg, iv, on days 1-4, 8-11of each 28 day cycle)
  After received induction therapy, patients will proceed to receive ASCT based on the willing of the patients and the decision of the investigators.
  Other Names: Induction Therapy (4 cycles); ASCT

SUMMARY:
This is a multicentre; single arm study in subjects with newly diagnosed multiple myeloma.

The primary objectives of this study is to assess the effect of bortezomib combination therapy (PAD regimen) followed by ASCT on bone metabolites in patients with newly diagnosed multiple myeloma, as measured by ELISA methodology as previously described analyzing the change in biochemical bone marker compared with the baseline value: bone formation marker- bone alkaline phosphatase(bALP) and osteoblast inhibitor- Dickkopf-1(DKK-1）.

The secondary objectives of this study are:

1. Subgroup analysis for the change from baseline in biochemical bone marker based on whether or not Bisphosphonate was used.
2. Assessment of other bone markers parameters: bone formation marker -carboxy terminal propeptide of type I procollagen (PICP); bone resorption markers -carboxy terminal telopeptide region of type I collagen ( ICTP); osteoclast stimulators -osteoprotegerin(OPG), soluble receptor activator of nuclear factor kappaB ligand(sRANKL);
3. To observe the effect of bortezomib on bone mineral density (BMD) as measured by repeated quantitative CT-scan;
4. The evaluation of Skeletal related events (SRE) and appearance of new bone lesions;
5. To determine progression free survival (PFS), 1 year survival, overall survival and safety profile following treatment with PAD and ASCT as first-line therapy.

DETAILED DESCRIPTION:
After providing written informed consent, subjects will be evaluated for eligibility during a 14-day screening period. Eligible subjects will receive 4 cycles PAD treatment prior to ASCT. Bisphosphonate therapy can be administered as medically indicated and according to local practice.

After the end of the treatment phase, there will be 18 months follow-up period for every patient with visits at 4, 6, 12 and 18 months after the end of the treatment phase. In case the disease progresses before completing the 18 months of follow-up and once the subject started alternative MM treatment, study assessments will stop, except for survival follow-up which will be collected every 6 months by either a telephone call or a visit to the study site. The follow-up for survival will continue for all subjects until the last subject has completed follow-up. One interim analysis of efficacy and safety will be performed when all subjects have achieved the end of treatment. Safety will be assessed by the monitoring of adverse events, physical examination, vital signs measurements and clinical laboratory tests.

ELIGIBILITY:
Inclusion Criteria:

1. Man or woman aged 18 to 65 years old;
2. Subjects are newly diagnosed MM patients which are scheduled by the investigators to be treated with vincristine, adriamycin and dexamethasone standard therapy. Stage II/III (according to Durie and Salmon criteria) with skeletal involvement, such as bone pain, bone lytic lesions, diffuse osteoporosis or pathologic fractures;
3. Life expectancy > 3 months;
4. Patient has measurable disease in which to capture response, defined as one or more of the following;

   * Serum M-protein level >10.0 g/L measured by serum protein electrophoresis or immunoglobulin electrophoresis; or
   * Urinary M-protein excretion > 1 g/24 hours; or
   * Bone marrow plasmacytosis of > 30% by bone marrow aspirate and/or biopsy; or
   * Serum free light chains (by the Freelite test) > 2 X the upper limit of normal (ULN), in the absence of renal failure.
5. Performance status (PS) of ECOG ≤2.0, unless PS of 3-4 based solely on bone pain;
6. Patients must have a Platelets count≥50×109 cells /L; Absolute neutrophil count (ANC)≥0.75×109 cells /L;
7. Patients must have adequate hepatic function defined as Alanine transaminase(ALT) ≤ 2.5 × upper limit of normal(ULN); Aspartate transaminase (AST) ≤2.5×ULN; Total bilirubin ≤2×ULN;
8. Patients must have adequate renal function defined as creatinine clearance >30 ml /min;
9. Subjects (or their legally acceptable representatives) must have signed a informed consent document indicating that they understand the purpose of and procedures required for the study and are willing to participate in the study.

Exclusion Criteria:

1. Non-secretory MM, unless the patient has measurable lesions on computed tomography (CT), magnetic resonance imaging (MRI) and/or positron emission tomography (PET);
2. Peripheral neuropathy or neuropathy pain grade 2 or high as defined by National Cancer Institute Common Terminology Criteria for Adverse Events(NCI CTCAE) Version 3;
3. Uncontrolled or severe cardiovascular disease, including myocardial infarction (MI ) within 6 months of enrollment, New York Heart Association (NYHA) Class III or IV heart failure, uncontrolled angina, clinically significant pericardial disease, or cardiac amyloidosis;
4. History of allergy reaction attributable to compounds containing boron or mannitol;
5. Any serious, active disease or psychiatric illness that could potentially interfere with the completion of treatment according to this protocol or the investigator's decision;
6. Concurrent treatment with another investigational agent;
7. Female subject who is pregnant or breast-feeding.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2012-12; Primary Completion 2016-09 (Actual); Study Completion 2017-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jian Hou, PhD, Principal Investigator — Shanghai Changzheng Hospital
Locations (1):
- Shanghai Changzheng Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- PAD Followed by ASCT: Drug: Bortezomib, Adriamycin (Doxorubicin) /Epidoxorubicin(EPI), Dexamethasone.
  After received induction therapy, patients will proceed to receive ASCT based on the willing of the patients and the decision of the investigators.
  PAD Followed by ASCT: Drug: Bortezomib, Bortezomib (1.3mg/m2, iv, on day 1, 4, 8, 11, of each 28 day cycle)
  Drug: Adriamycin (Doxorubicin) /EPI, Adriamycin (Doxorubicin) (9 mg/m2, iv, on days 1-4 of each 28 day cycle) or EPI (15mg/m2, iv, on days 1-4 of each 28 day cycle)
  Drug: Dexamethasone, Dexamethasone (20mg, iv, on days 1-4, 8-11of each 28 day cycle)
  After received induction therapy, patients will proceed to receive ASCT based on the willing of the patients and the decision of the investigators.
Period: Overall Study
Arm/Group | PAD Followed by ASCT
Started | 18
Completed | 0
Not Completed | 18

BASELINE CHARACTERISTICS:
Arm/Group | PAD Followed by ASCT
Number analyzed (Participants) | 18
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 18
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.1 (6.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 12
Region of Enrollment [Count of Participants; unit: Participants]
  China | 18

OUTCOME MEASURES:

1. Primary Outcome: Bone Formation Markers Measurement
Description: The bone formation marker- bone alkaline phosphatase(bALP) and osteoblast inhibitor- Dickkopf-1(DKK-1）are measured on serum samples by ELISA methodology at baseline, on day 28 of cycles 1,4, and after 4, 6, 12 and 18 months of follow-up or until start of alternative multiple myeloma(MM) treatment, if earlier.
Time Frame: Up to Cycle 4 with 28 days per cycle
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | PAD Followed by ASCT
Number analyzed (Participants) | 18
U/L
  bALP on baseline | 21.87 (14.11)
  bALP after cycle 1 | 23.2 (12.89)
  bALP changes from baseline to cycle 1 | 1.33 (1.02)
  bALP after cycle 4 | 28.75 (13.12)
  bALP changes from baseline to cycle 4 | 6.88 (3.20)
  DKK-1 on baseline | 4765 (159.5)
  DKK-1 aftercycle 1 | 2653 (135.2)
  DKK-1 changes from baseline to cycle 1 | 2653 (135.2)
  DKK-1 after cycle 4 | 1589 (128.2)
  DKK-1 changes from baseline to cycle 4 | 3176 (123.8)
Statistical Analysis 1: Comparison: PAD Followed by ASCT; bALP changes from baseline to cycle 1; Test type: Other; p = 0.002, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: PAD Followed by ASCT; b-ALP changes from baseline to cycle 4; Test type: Other; p < 0.001, t-test, 2 sided
Statistical Analysis 3: Comparison: PAD Followed by ASCT; DKK-1 changes from baseline to cycle 1; Test type: Other; p = 0.005, Wilcoxon (Mann-Whitney)
Statistical Analysis 4: Comparison: PAD Followed by ASCT; DKK-1 changes from baseline to cycle 4; Test type: Other; p < 0.001, t-test, 2 sided

2. Secondary Outcome: Measurement of Bone Mineral Density
Description: The effect on bone mineral density（BMD） will be measured by quantitative analysis of qCT scans of the intra-individual same region [lumbar spine and hip] at baseline, on day 28 of cycles 4, and after 4, 6, 12 and 18 months of follow-up or until start of alternative MM treatment, if earlier.
Time Frame: At baseline, on day 28 of cycles 1,4, and after 4, 6, 12 and 18 months of follow-up or until start of alternative MM treatment
Population: Data were not collected.
Arm/Group | PAD Followed by ASCT
Number analyzed (Participants) | 0

3. Secondary Outcome: Skeletal Related Events' Evaluation
Description: Skeletal survey of the skeleton using plain radiography will be performed at baseline, on day 28 of cycle 4, and after 6, 12 and 18 months of follow-up or until start of alternative MM treatment, if earlier. SREs, such as pathological fractures, need for radiation therapy or surgery will be recorded at the time of the event.
Time Frame: At baseline, on day 28 of cycles 4, and after 4, 6, 12 and 18 months of follow-up or until start of alternative MM treatment
Population: Data were not collected.
Arm/Group | PAD Followed by ASCT
Number analyzed (Participants) | 0

4. Other Pre Specified Outcome: Evaluation of Responses
Description: Evaluation of responses was performed every cycle. Responses were assessed according to the european group for blood and marrow transplantation（EBMT） criteria (An attempt will be made to collect data for the assessment of stringent complete response (sCR) if these data are available.). Other efficacy parameters including PFS and 1-year overall survival rate and overall survival will be evaluated by normal methodology. According to EBMT criteria, responses were assessed by changes in the level of the serum paraprotein and/or urinary light chain excretion.The specific assessment rules may refer to EBMT criteria for MM.
Time Frame: At baseline, on day 28 of cycles 4, and after 4, 6, 12 and 18 months of follow-up
Measure: Count of Participants; unit: Participants
Arm/Group | PAD Followed by ASCT
Number analyzed (Participants) | 18
Participants
  After 4-month PAD treatment: sCR | 4
  After 4-month PAD treatment: CR | 0
  After 4-month PAD treatment: PR | 12
  After 4-month PAD treatment: MR | 1
  After 4-month PAD treatment: NC | 1
  After 4-month PAD treatment: PD | 0
  After ASCT: sCR | 4
  After ASCT: CR | 0
  After ASCT: PR | 12
  After ASCT: MR | 1
  After ASCT: NC | 1
  After ASCT: PD | 0
  End of study: sCR | 2
  End of study: CR | 1
  End of study: PR | 9
  End of study: MR | 1
  End of study: NC | 1
  End of study: PD | 4

5. Other Pre Specified Outcome: Safety Evaluation
Description: Safety evaluations will be based on scheduled physical examinations, Eastern Cooperative Oncology Group(ECOG) scores, vital signs (blood pressure, heart rate) and clinical laboratory tests.
Time Frame: Starting with informed consent signature through study completion, an average of 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | PAD Followed by ASCT
Number analyzed (Participants) | 18
Participants
  AE | 15
  TEAE | 15
  TEAE related to treatment | 14
  TEAE(CTCAE≥3) | 11
  TEAE related to treatment(CTCAE≥3) | 10
  SAE | 0

6. Other Pre Specified Outcome: Evaluation of Responses(PFS)
Description: Efficacy parameters PFS will be evaluated by normal methodology. PFS =（date of signing informed consent form minus the date of first documented progression or date of death from any cause plus 1）/30.5（months）
Time Frame: From date of signing informed consent form until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 100 months
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | PAD Followed by ASCT
Number analyzed (Participants) | 18
months | 13.7 [10.3 to 13.7]

ADVERSE EVENTS:
Time Frame: On baseline, on day 28 of cycles 1,4, and after 4, 6, 12 and 18 months of follow-up or until start of alternative MM treatment
Arm/Group | PAD Followed by ASCT
All-Cause Mortality (participants affected / at risk) | 0/18
Serious Adverse Events (participants affected / at risk) | 0/18
Other Adverse Events (participants affected / at risk) | 15/18
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PAD Followed by ASCT (N=18)
ALT rise (Hepatobiliary disorders) | 1 (1)
Herpes zoster (Infections and infestations) | 3 (3)
Leukopenia (Blood and lymphatic system disorders) | 8 (14)
Perineural inflammation (Infections and infestations) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 7 (19)
Constipation (Gastrointestinal disorders) | 2 (3)
Hypokalemia (Blood and lymphatic system disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 3 (3)
Fever (General disorders) | 3 (4)
Hypodynamia (General disorders) | 1 (1)
Pulmonary infection (Infections and infestations) | 1 (4)
Diarrhea (Gastrointestinal disorders) | 3 (3)
Hyperbilirubinemia (Blood and lymphatic system disorders) | 1 (1)
Hyperuricemia (Blood and lymphatic system disorders) | 1 (1)
Lymphopenia (Blood and lymphatic system disorders) | 3 (4)
Hypoalbuminemia (Blood and lymphatic system disorders) | 2 (2)
Vomiting (Gastrointestinal disorders) | 2 (2)
Rash (General disorders) | 1 (1)
Edema (General disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No